CLINICAL TRIAL: NCT02132286
Title: Serotonin Transporter Genetic Variation and Amygdala Responses to Quetiapine and Selective Serotonin Reuptake Inhibitor Treatment in Major Depression
Brief Title: Serotonin Transporter Genetic Variation and Amygdala Responses to Antidepressant Medications in Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Rajamannar Ramasubbu, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: D1443L00037
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder
Keywords: Functional magnetic resonance neuroimaging; Serotonin transporter gene polymorphism; Amygdala; Antidepressant; Quetiapine; Citalopram; imaging biomarker
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine -XR (extended release) (Experimental): Quetiapine-XR (extended release) 150-300mg- treatment in MDD patients with S/Lg alleles in MDD
  Interventions: Drug: Quetiapine XR (extended release)
- Citalopram (Active Comparator): Citalopram 10-20 mgm/day treatment for 8 weeks in MDD with S/Lg alleles
  Interventions: Drug: Quetiapine XR (extended release)

INTERVENTIONS:
Drug: Quetiapine XR (extended release) — Treatment of quetiapine XR ( extended release)in MDD patients with S/Lg alleles
  Other Names: Seroquel XR (extended release)

SUMMARY:
Major depressive disorder (MDD) is a highly prevalent, chronic and/or recurrent condition with substantial morbidity and mortality. It is one of the leading causes of disability worldwide. Despite significant advances in pharmacological treatment for depression over the last two decades, a significant proportion of patients (10-20%) are resistant to currently available treatment. The development of new effective treatment for depression is limited by the fact that MDD is a heterogeneous disorder with subgroups based on variations in etiological factors and treatment response. Functional magnetic resonance imaging (fMRI) approaches offer promise in the prediction and evaluation of clinical response of antidepressant treatment.

Previous fMRI studies have identified increased activity in dorso-lateral prefrontal cortex (DLPFC) and decreased amygdala activity from the baseline as imaging markers of antidepressant response in patients with MDD. However, these studies have examined MDD as a homogenous group without specifying the type of patient group, and brain regions as a priori hypothesis.We therefore need studies using combined genetics and neuroimaging measures as biomarkers in the prediction and evaluation of clinical response to antidepressants. In this study we attempted to determine imaging clinical efficacy markers in previously defined brain regions (amygdala and prefrontal regions) for two classes of antidepressants (citalopram and quetiapine extended release (XR)) with differential action on serotonin transporter inhibition in a subgroup of MDD patients with high risk allele ( S/Lg) of serotonin transporter gene polymorphism.

DETAILED DESCRIPTION:
Background

The atypical antipsychotic quetiapine has been found to have significant antidepressant action in addition to antipsychotic action. Unlike citalopram a selective serotonin reuptake inhibitor (SSRI) quetiapine has no effect on serotonin transporter (5-HTT) but it increases post synaptic 5-HT1A binding potentials and down regulates 5-HT2A receptors consistently (Tarazi et al., 2002) due to its direct antagonistic effect on 5-HT2A receptors and agonistic effect on post synaptic 5-HT1A receptors. The quetiapine induced down regulation of 5-HT2A receptors and increased density of 5-HT1A receptors has been attributed to its antidepressant effects (Thase et al., 2006). Taking into account that contrary to SSRIs, quetiapine mediated antidepressant effect does not depend on 5-HTT inhibition, it is possible that genetic factors which regulate 5-HTT expression may have less influence on the outcome of quetiapine treatment than on SSRI treatment in depressed patients.

Rationale for this study

In this experiment, we proposed to study the efficacy of quetiapine relative to citalopram in patients with MDD and high risk serotonin transporter gene polymorphism (5-HTTLPR)S/Lg alleles. Since 5-HTTLPR-S/Lg allele confers vulnerability to depression in the context of emotional stress (Caspi et al., 2003) and also mediates poor and slower response to SSRI antidepressants (Serretti et al., 2007), a study of this nature will have significant treatment implications in depressed patients with high risk for stress induced relapses and treatment resistance. Given that quetiapine has no affinity for 5-HTT and may normalize the receptor changes that occur in conditions with low 5-HTT expression (S and Lg carriers and patients with MDD), we predict that compared to citalopram treatment, quetiapine treatment will be more effective in reducing amygdala responses to negative stimuli as well as depressive symptoms in patients with MDD and high risk S/Lg alleles. It is also predicted that because of its direct action on post synaptic 5-HT1A and 5-HT2A receptors, quetiapine treatment will show early onset of action on amygdala responses than citalopram treatment especially in patients with S allele.

Primary Hypothesis: There will be a significant decrease in amygdala responses to negative facial stimuli in depressed patients with S/Lg allele after short term (1 week) and long term (8 weeks) quetiapine treatment compared to citalopram treatment.

Secondary Hypotheses: The reduction in amygdala responses at week 8 of treatment will correlate with clinical improvement, and the reduction in amygdala responses at week one of the treatment may predict the subsequent clinical response at week 8.

Study Objective

To examine the effects of short term (1 week) and long term (8 weeks) treatment of quetiapine 150-300 mg and citalopram 10-20 mg on amygdala responses to negative emotional stimuli in patients with major depression with high risk alleles (S/Lg)

Study Plan and Procedures

This is an eight-week, parallel-group, randomized, double blind comparative trial with a repeated measure design in which the patients with major depression will be randomly assigned in a 1:1 ratio to receive treatment with either quetiapine 300 mg or citalopram 20mg for an 8-week period. The subjects will undergo imaging during three separate 60-minute sessions: 1) baseline or week 0, 2) one week after initiation of treatment, and 3) 8 weeks after baseline or initiation of treatment. Genotyping will be performed in all participants.

64 Caucasians of both gender with an age range of 20-55 years meeting the criteria of DSM-IV (American Psychiatric Association 2000) criteria for major depressive disorder according to the Structured Clinical Interview (First et al.,2000) for DSM-IV Axis 1 disorders will be recruited from the Calgary Health Region outpatient mental health clinics and through local newspaper advertisements. Eligible patients will be randomly assigned in a 1:1 ratio to receive either quetiapine or citalopram. Thus each treatment arm will have 32 subjects.

Clinical assessment and treatment

At the baseline, Structured Clinical Interview I and II will be performed to determine the DSM IV diagnosis of MDD and also to exclude other Axis I psychiatric disorders. Hamilton rating scale for depression (HRSD) (will be used to assess the severity of depressive symptoms (Hamilton 1960) and Hamilton anxiety rating scale (HAM-A) (Hamilton 1959) will be used to rate anxiety symptoms. Additionally, temperament and character inventory (TPI) (Cloninger et al 1994) and childhood trauma questionnaire (CTQ) will be administered to assess and control for the personality traits such as fear and anxiety and child hood abuse that are known to affect amygdala responses to fearful stimuli

After the baseline assessment and prior to the initiation of treatment, first fMRI session will be performed. Then quetiapine XR will be initiated at 50mg/day the first 2 days and 150 mg/day on day 3 and titrated to 300mg/day by day 4, and citalopram will be initiated at the dose of 10 mg /day and titrated to 20 mg/day by day 4. The patients in both treatment arms will continue this dosage until the completion of the study protocol 8 weeks later. For the patients who could not tolerate or develop adverse effects, the quetiapine dose will be reduced to 150 mg/day and citalopram dose will be reduced to 10 mg/day. The patients who could not tolerate quetipine 150 mg/day and citalopram 10 mg/day will be terminated from the study.During their participation in the study, patients will undergo a clinical assessment at week one after the titration of quetiapine and citalopram and a second fMRI session. Depressive and anxiety symptoms will be rated using HRSD and HAM-A. Then, patients will be evaluated every two weeks and at the week 8 using HRSD and HAM-A. At week 8, a third fMRI session will be performed. Adverse effects will be recorded. The patients who could not tolerate any of the study medications will be terminated from the study

Genotyping

Genotyping of 5-HTTLPR and functional single nucleotide polymorphism (SNP)(A-G) rs 25531 at the promoter region will be performed using polymerase chain reaction (PCR) followed by double restriction endonuclease digestion as reported previously (Wendland et al., 2006) . High resolution agarose gel will be used to determine four alleles: Sa-469 bp (uncut), Sg-402+67 bp, La- 512 bp (uncut), and Lg-402+110bp.

fMRI

fMRI will be performed on three occasions: i) at the baseline, ii) 1 week after optimizing the treatment, iii) 8 weeks after optimization An fMRI block design with presentations of angry and fearful facial expressions interleaved with a sensorimotor control task will be used to elicit activations in amygdala. This paradigm of perceptual processing of facial expressions of negative emotions has been shown to effectively and consistently activate amygdala in previous studies (Hariri et al., 2002). The paradigm consists of a total of 6 runs and during each run, 3 blocks of emotional task interleaved with 4 blocks of sensorimotor control task will be presented. During the emotion task, subject will view a trio of faces and select one of two faces that expresses the same emotion as the target face in the top. Each emotion block will consist of 6 images, three of each gender, and target affect (angry and fear). Each facial stimulus will be presented for 5 seconds. The identity of all three faces will be always different. During the sensorimotor control task, subjects will view a trio of geometric shapes (circles, vertical and horizontal ellipses) and select one of two shapes that matches the target shape. Each control block consists of 6 different images, and each image will presented for 5 seconds. Accuracy and reaction time will be recorded during all scans.

Method of statistical analysis

The first level of analysis will be the generation of fMRI maps of brain activity using FMRIB Software Library (FSL), a statistical software package specifically designed for fMRI applications, which uses the general linear model to compute contrast parameter estimates of explanatory variables (in our case, the explanatory variable is face task vs. sensorimotor task) for each pixel in the brain images. The result is an estimate of the response magnitude in a given pixel that surpasses a specified statistical threshold (typically, p = 0.01).

The main variable of interest will be the magnitude of activity within the amydala. For each patient, regions of interest (ROIs) will be drawn manually to encompass the amygdala within each hemisphere with the aid of each patient's anatomical images. Magnitude of activity with the ROIs will be recorded. A generalized linear mixed model will be used to analyze group data with treatment, and time of session (baseline, 1-week, 8-week) as factors into the analysis. As we expect that the sample size of patients with La/La genotype will be smaller in each treatment group, the primary analysis will be done only in MDD patients with S/Lg alleles to prove our hypothesis. To examine the association between changes in amygdala activity and response in depression severity the change in HAM-D for each patient over 8 weeks will be regressed on the corresponding change in amygdala activity. A similar approach will be used to correlate 1-week change in activity with 8-week change in depression severity. The other regions that are functionally or structurally connected with amygdala such as anterior cingulate region (ACC), dorso-lateral prefrontal cortex (DLPFC), dorso-medial prefrontal cortex (DMPFC), and precuneus (PCC) will also be selected for exploratory analysis

The potential confounding factors such as age,sex, childhood adversity and personality index of fear and anxiety, baseline depression and anxiety scores will be controlled between the groups or will be covaried if there are intergroup differences in these variables.

Determination of sample size

As it is expected that approximately 70% of participants will express the S/Lg allele, the magnitude of activity within the amygdala is estimated from a meta-analysis by Munafo et al (2008). to be 0.10 with a standard deviation of 0.11 Assuming a difference in mean change (baseline to 8 weeks) between groups to be 0.05 with a change standard deviation of 0.07, a total of 32 patients per group is required to detect this difference with 80% power at a two-sided 5% level of significance. A 50% difference in mean change is reasonable based upon the results by Sheline et al (2001).

ELIGIBILITY:
Inclusion Criteria

1. A diagnosis of Major Depressive Disorder of unipolar subtype by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) and a score of 18 on the 17-item Hamilton Rating Scale for Depression (HRSD) (Hamilton 1960).
2. Both females and males aged 18 to 65 years of Caucasian descent.The association between 5-HTTLPR- s allele and poor response to SSRIs is significant only in Caucasians
3. Female patients of childbearing potential must be using a acceptable method of contraception ( contraceptive pill, injection or patch, vaginal ring, intra-uterine device, female condom, contraceptive sponge, diaphragm, cervical cap, lea contraceptive, tubal ligation, natural birth control methods, and withdrawl) and have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
4. Able to understand and comply with the requirements of the study 5 All participants should be free of psychotropic medication for a minimum of 4 weeks at recruitment

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria.
3. Major depression with mood congruent and incongruent psychotic symptoms
4. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
5. Known intolerance or lack of response to quetiapine fumarate and citalopram as judged by the investigator
6. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
7. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
8. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
9. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
10. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment will be excluded. However, patient with occasional use of above mentioned substance but does not fulfil abuse criteria according to DSM-IV during the defined period will be included in the study.
11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
12. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
13. Involvement in the planning and conduct of the study
14. Previous enrolment or randomisation of treatment in the present study.
15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
16. A patient with unstable Diabetes Mellitus (DM) 17 Subjects who are contraindicated for MRI (pregnancy, metal implants) will be excluded.

18. Severe claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes in amygdala responses to negative emotional faces from the pre-treatment baseline to 8 weeks post treatment. | 8 weeks
  Consistent with the hypothesis of this study, the primary outcome variable will be the magnitude of Blood Oxygen Level Dependent Responses ( BOLD) within the amygdala as measured by changes in amygdala activation from baseline at week 8 of the treatment in the two treatment groups.

SECONDARY OUTCOMES:
Changes in depression symptom severity as measured by Hamilton Depression Rating Scale from the pre-treatment baseline to week 8 post-treatment | 8 weeks
  This clinical efficacy secondary outcome measure is required to correlate with primary measure of amygdala responses to determine whether amygdala changes will be a clinical efficacy surrogate imaging marker.

OTHER OUTCOMES:
changes in activity in cingulate and prefrontal regions from the baseline to 8 weeks post treatment | 8 weeks
  These regions are functionally connected with amygdala and also have shown changes with antidepressant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rajamannar Ramasubbu, MD, FRCPC., Principal Investigator — University of Calgary
Locations (1):
- University of Calgary: Foothills medical centre, Calgary, Alberta, Canada